CLINICAL TRIAL: NCT04742309
Title: A Randomized, Subject-Masked, Active-Controlled, Parallel-Arm Clinical Trial Comparing Pecs-2 and Paravertebral Nerve Blocks
Brief Title: Pectoralis Block vs Paravertebral Nerve Blocks for Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pecs vs PVB
Record Dates: First submitted 2021-01-29; First posted 2021-02-08 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Breast Surgery
Keywords: Regional Anesthesia; Pecs-2; Paravertebral nerve block
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Anesthesia teams in the operating rooms and recovery room nurses will be masked to treatment group assignment (therefore, the primary outcome measure collection). Outcomes assessor for the questionnaire involving secondary outcomes on the day following surgery will not be masked to treatment group, although subjects will remain masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pecs-2 (Experimental): For Pecs-2 blocks, the needle will be advanced to the tissue plane between the pectoralis major and minor muscles at the vicinity of the pectoral branch of the acromiothoracic artery where 10 mL of local anesthetic will be deposited. In a similar manner, 20 mL will be deposited at the level of the third rib above the serratus anterior muscle with the intent of spreading injectate to the axilla. The study fluid will be ropivacaine 0.3% with epinephrine.
  Interventions: Drug: Pecs-2 block (single injection)
- Paravertebral (Active Comparator): For paravertebral blocks, ropivacaine 0.5% (with epinephrine) 9 mL will be administered at each of two levels per side: the T3 and T5 levels for sides without axillary involvement; and at the T2 and T4 level for sides with axillary involvement.
  Interventions: Drug: Paravertebral block (single injection)

INTERVENTIONS:
Drug: Pecs-2 block (single injection) — For Pecs-2 blocks, the needle will be advanced to the tissue plane between the pectoralis major and minor muscles at the vicinity of the pectoral branch of the acromiothoracic artery where 10 mL of local anesthetic will be deposited. In a similar manner, 20 mL will be deposited at the level of the third rib above the serratus anterior muscle with the intent of spreading injectate to the axilla. The study fluid will be ropivacaine 0.3% with epinephrine.
  Arms: Pecs-2
Drug: Paravertebral block (single injection) — For paravertebral blocks, ropivacaine 0.5% (with epinephrine) 9 mL will be administered at each of two levels per side: the T3 and T5 levels for sides without axillary involvement; and at the T2 and T4 level for sides with axillary involvement.
  Arms: Paravertebral

SUMMARY:
Following painful surgical procedures of the breast, postoperative analgesia is often provided with a nerve block called a "paravertebral" block. For intense, but shorter-duration acute pain, a single-injection of numbing medicine is used which lasts about 12 hours. Recently, a new type of block has been reported: the "Pecs-2" block. The theoretical benefits include ease of administration since it is closer to the skin (less deep) compared with the paravertebral block and therefore easier to identify and target with ultrasound (therefore increasing success rate); and, a lower risk of complications. Lastly, it might be easier to insert a tiny tube which would allow additional numbing medicine to be injected. There are, therefore, multiple theoretical reasons to prefer the Pecs-2 over the paravertebral nerve block. Unfortunately, it remains unknown if the pain control provided by this new type of block is comparable to that provided with the older block. The investigators therefore propose to compare these two blocks with a clinical study.

DETAILED DESCRIPTION:
This investigation will be a randomized, subject-masked, active-controlled parallel-arm, human subjects clinical trial. Of note, the investigators will be using standard-of-care local anesthetic under a Food and Drug Administration-approved purpose and do not plan to research a possible change of indication or use of these medications as part of this research project. The treatments in both groups are currently used at our institution and there is true clinical equipoise at this time. The only difference in treatment between subjects who enroll versus those not enrolled in this study will be those who enroll will have the decision between which anatomic block location determined randomly, as opposed to the physician simply choosing him/herself.

Enrollment. Consenting adults undergoing breast surgery with a planned single-injection regional analgesic will be offered enrollment. Patients undergoing breast surgery with a planned perineural catheter regional analgesic will be excluded. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current University of California San Diego Institutional Review Board-approved informed consent form. Selection for inclusion will not be based on gender, race, or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status.

Preoperative Procedures. Following written, informed consent, the investigators will collect baseline anthropomorphic information (e.g., age, sex, height, and weight). All subjects will have a peripheral intravenous catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and placed in the sitting position. Intravenous midazolam and fentanyl will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. Both possible block locations will be viewed with ultrasound. If one or both of the locations is unacceptable for block placement in the clinician's opinion, the subject will not be randomized and will not proceed further with the study.

Subjects will then be randomized using a computer-generated list and opaque, sealed envelopes to one of two treatment groups: (blocks of 4, stratified for unilateral vs. bilateral surgery): (1) Pecs-2 or (2) paravertebral block. All blocks will be placed by a regional anesthesia fellow or resident under the direct supervision and guidance of a regional anesthesia attending (or by the attending themselves).

For paravertebral blocks, a total of 18 mL of ropivacaine 0.5% with epinephrine will be administered per side (90 mg). An equivalent mass of ropivacaine will be administered for the Pecs-2 blocks (90 mg), but since more volume is required (30 mL per treated side), the concentration will be decreased to 0.3% ropivacaine (with epinephrine). Therefore, for bilateral procedures, 90 mg will be administered to each side (180 mg total, with epinephrine). The area of needle insertion will be cleaned with chlorhexidine gluconate and isopropyl alcohol. All blocks will be placed using standard UCSD ultrasound-guided techniques as previously described.

For Pecs-2 blocks, the needle will be advanced to the tissue plane between the pectoralis major and minor muscles at the vicinity of the pectoral branch of the acromiothoracic artery where 10 mL of local anesthetic will be deposited. In a similar manner, 20 mL will be deposited at the level of the third rib above the serratus anterior muscle with the intent of spreading injectate to the axilla.

For paravertebral blocks, ropivacaine 0.5% 9 mL will be administered at each of two levels per side: the T3 and T5 levels for sides without axillary involvement; and at the T2 and T4 level for sides with axillary involvement.

Single-injection blocks will be considered successful if, within 30 minutes, the subject experiences decreased sensation to cold temperature with an alcohol pad over the approximate level of the ipsilateral 4th thoracic dermatome. Misplaced blocks will be replaced successfully, or the patient excluded from further study participation. For subjects undergoing bilateral surgical procedures, a block using the same protocol will be administered on the contralateral side.

Intraoperatively, all subjects will receive a general anesthetic using inhaled and intravenous anesthetic and oxygen. Intravenous fentanyl will be administered for cardiovascular responsiveness to noxious stimuli at the discretion of the anesthesia provider.

Postoperatively: Subjects will be discharged with a prescription for oxycodone 5 mg tablets for supplementary analgesia and instructed to record the time at which they take their first opioid tablet as well as the time at which they believe the block starts to wear off.

Outcome measurements (end points). Pain scores will be recorded using the Numeric Rating Scale. Within the recovery room, pain scores, opioid requirements, and antiemetic administration will be recorded by nursing staff masked to treatment group. The morning following surgery, all subjects will be contacted by phone or in person [if hospitalized] to record lowest, average, highest, and current pain scores; sleep disturbances, and nausea using a 0-10 Likert scale (0 = no nausea; 10 = vomiting). For outpatients, opioid requirements will be recorded while inpatients will have opioid requirements extracted from the electronic medical record. In addition, the investigators will extract antiemetic use from the electronic record. The investigators will collect the times at which subjects felt their block resolve and they consumed their first opioid analgesic pills following recovery room discharge.

Hypothesis 1: Following breast surgery, analgesia will be non-inferior in the recovery room with a Pecs-2 block compared with a paravertebral block as measured with the Numeric Rating Scale.

Hypothesis 2: For breast surgery, opioid consumption will be non-inferior in the operating and recovery rooms with a Pecs-2 block compared with a paravertebral block (primary: cumulative intravenous morphine equivalents).

Primary end point: In order to claim that Pecs-2 blocks are non-inferior to paravertebral blocks, both Hypotheses 1 and 2 must be at least non-inferior.

Statistical methods. Descriptive statistics will be provided by arm and in aggregate. Baseline characteristics of arms will be compared using the Wilcoxon-Mann-Whitney and Fisher's Exact tests. Key characteristics that are significantly different (p<0.05) will be included as covariates in the analysis models.

Primary aim. The investigators will test the noninferiority of the Pecs-2 nerve block compared to the paravertebral nerve block. The 95% confidence interval (CI) associated with the Wilcoxon-Mann-Whitney test will be derived for the group difference (paravertebral minus serratus) in median pain scores within the recovery room. If the lower limit of the 95% CI is greater than -1.25, the investigators will conclude noninferiority. If there are significant differences between the groups in any key characteristics, these characteristics will be included as covariates in a linear model. The same noninferiority margin (-1.25) will be applied to the 95% CI for the covariate adjusted group difference in mean pain derived from the linear model.

The noninferiority of the Pecs-2 nerve block with regard to total opioid consumption within the operating and recovery rooms will be tested in the same manner as pain, i.e. comparing the limits of a 95% confidence interval associated with the Wilcoxon-Mann-Whitney test to a predefined noninferiority margin (in this case 2 mg). Covariate adjusted linear models will again be applied in the event that key characteristics are significantly different between the groups.

Sample size justification. Power for the Wilcoxon-Mann-Whitney derived noninferiority testing is based on 10,000 simulated trials. The investigators simulated pain scores from a discrete distribution with median of 3 (interquartile range of 2-5). Between the quartiles, the probability of each score was assumed constant. The distribution for each group was assumed to be the same. The sample size of n=50 per group provides 82% power to detect noninferiority in pain with a margin of 1.25. Similarly, opioid consumption was assumed to follow a truncated normal distribution with mean 2.5 mg and standard deviation 2 mg, and minimum value 0 mg. The sample size of n = 50 per group provides at least 95% power to detect noninferiority with margin 2 mg. However, the investigators will increase the number of enrolled subjects to account for an unanticipated higher variability for both outcomes. Therefore, the investigators will enroll 75 subjects for each of two treatments with primary end point values for a total enrollment of 150 subjects with a primary end point. To allow for dropouts, the investigators request a maximum enrollment of 175 subjects. Noninferiority in pain is tested first, and if significant, noninferiority in opioid consumption is tested. Under this hierarchical testing framework, no adjustment in alpha is necessary to control Type 1 error.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing unilateral or bilateral breast surgery with at least moderate postoperative pain anticipated.
2. Analgesic plan includes a single-injection peripheral nerve block(s).
3. Age 18 years or older.

Exclusion Criteria:

1. Morbid obesity as defined by a body mass index > 40 (BMI=weight in kg / [height in meters]2).
2. Renal insufficiency ( abnormal preoperative creatinine or eGFR)
3. Chronic opioid use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks).
4. History of opioid abuse.
5. Any comorbidity which results in moderate or severe functional limitation inability to communicate with the investigators or hospital staff.
6. Inability to communicate with the investigators or hospital staff.
7. Pregnancy
8. Planned regional analgesic with perineural catheter placement
9. Incarceration
10. Known allergy to amide local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD,MS, Principal Investigator — UCSD Medical Center
Locations (1):
- University Of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pecs-2 | Paravertebral
Started | 60 | 59
Completed | 60 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pecs-2 | Paravertebral | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (15) | 45 (16) | 50 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119
Height (cm) [Mean (Standard Deviation); unit: cm] | 165 (8) | 165 (8) | 165 (8)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 70 (15) | 70 (14) | 70 (15)
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kg /m^2] | 25.6 (4.9) | 25.7 (5.1) | 25.6 (5.0)
Bilateral procedure (%) [Count of Participants; unit: Participants] | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Recovery Room Numeric Rating Scale Pain Scores
Description: Numeric Rating Scale: the NRS is a segmented numeric version of the Visual Analog Scale (VAS) in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes. Of note, in order to claim that Pecs-2 blocks are non-inferior to paravertebral blocks, both Hypotheses 1 and 2 must be at least non-inferior.
Time Frame: From arrival in the recovery room until recovery room discharge, assessed up to 12 hours total
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
score on a scale | 3.3 [2.3 to 4.8] | 1.3 [0 to 3.6]

2. Primary Outcome: Cumulative Operating and Recovery Room Opioid Consumption
Description: The morphine equivalents consumed in both the operating and recovery rooms. Of note, in order to claim that Pecs-2 blocks are non-inferior to paravertebral blocks, both Hypotheses 1 and 2 must be at least non-inferior.
Time Frame: From entering the operating room until recovery room discharge, assessed up to 24 hours
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
mg | 18 [13 to 22] | 10 [10 to 20]

3. Secondary Outcome: Nausea and Vomiting
Description: 0-10 Likert scale (0 = no nausea; 10 = vomiting)
Time Frame: Recovery room discharge until data collection call on Postoperative Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
score on a scale | 0.1 (0.3) | 0.1 (0.3)

4. Secondary Outcome: Time of First Opioid Use
Description: We attempted to collect the times at which participants identified block resolution and their first oral opioid analgesic following recovery room discharge. However, the majority of participants could not recall this information with confidence, and we therefore ceased attempting to collect this data. There is no data to present.
Time Frame: Recovery room discharge until data collection call on Postoperative Day 1
Population: We attempted to collect the times at which participants identified block resolution and their first oral opioid analgesic following recovery room discharge. However, the majority of participants could not recall this information with confidence, and we therefore ceased attempting to collect this data.
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time of Block Resolution
Description: as for outcome 4
Time Frame: Recovery room discharge until data collection call on Postoperative Day 1
Population: as for outcome 4
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Opioid (Oxycodone) Consumption
Description: The amount of a synthetic opioid, oxycodone, that was consumed during the time period measured in oxycodone equivalents
Time Frame: Recovery room discharge until data collection call on Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
mg | 5 [5 to 10] | 5 [0 to 10]

7. Secondary Outcome: Worst Pain Measured Using the Numeric Rating Scale Pain Score
Description: Numeric Rating Scale: the Numeric Rating Scale is a segmented numeric version of the Visual Analog Scale in which the study subject selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. This 11-point numeric scale ranges from 0 representing "no pain" to 10 representing "worst imaginable pain." Higher numeric scores represent increased pain and thus worse outcomes.
Time Frame: Recovery room discharge until data collection call on Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
score on a scale | 5 [3.8 to 6.0] | 3 [2 to 5]

8. Secondary Outcome: Lowest Pain Measured Using the Numeric Rating Scale Pain Score
Description: as for outcome 7
Time Frame: Recovery room discharge until data collection call on Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
score on a scale | 3 [0 to 3] | 0 [0 to 2]

9. Secondary Outcome: Average Pain Measured Using the Numeric Rating Scale Pain Score
Description: as for outcome 7
Time Frame: Recovery room discharge until data collection call on Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
score on a scale | 3 [2 to 4] | 1.8 [0 to 3]

10. Secondary Outcome: Current Pain Measured Using the Numeric Rating Scale Pain Score
Description: as for outcome 7
Time Frame: Postoperative Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
score on a scale | 2 [2 to 3] | 1 [0 to 2]

11. Secondary Outcome: Awakenings Due to Pain
Description: The number of times subject recalls awakening from sleep due to pain
Time Frame: Evening of surgery
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Pecs-2 | Paravertebral
Number analyzed (Participants) | 60 | 59
episodes | 0.2 (0.4) | 0.2 (0.4)

ADVERSE EVENTS:
Time Frame: From enrollment preoperatively through the day following surgery (approximately 24 hours)
Arm/Group | Pecs-2 | Paravertebral
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 0/60 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04742309/Prot_SAP_000.pdf